CLINICAL TRIAL: NCT06425211
Title: Effectiveness of Pelvic Floor Therapy for the Management of Erectile Dysfunction and Premature Ejaculation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMGC-6
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Erectile Dysfunction; Premature (Early) Ejaculation; Premature Ejaculation; Pelvic Floor; Weak
MeSH Terms: conditions — Erectile Dysfunction; Premature Birth; Premature Ejaculation; Asthenia | interventions — Exercise Therapy; Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Erectile Dysfunction (Experimental): The therapy depends if patient is classified within muscular hyperactivity or muscular hypoactivity.
  For muscular hypoactivity:
  Pelvic Floor Physiotherapy assessment: session 1 Proprioceptive and Coordination Work: sessions 2-7 Muscle workout: sessions 8-15 Functional training: sessions 16-23 Final evaluation: Session 24
  For muscular hyperactivity they will be given:
  Pelvic Floor Physiotherapy assessment: session 1 Proprioceptive and Coordination Work: sessions 2-7 Muscle workout: sessions 8-15 Functional training: sessions 16-23 Final evaluation: session 24
  These interventions include: Therapeutic exercises, Perineal electromyographic biofeedback, and Electrical stimulation
  Interventions: Behavioral: Therapeutic exercises; Device: Perineal electromyographic biofeedback; Device: Electrical stimulation
- Premature Ejaculation (Experimental): Pelvic Floor Physiotherapy assessment: session 1 Proprioceptive and Coordination Work: sessions 2-15 Muscle workout: sessions 16-19 Functional training: sessions 20-23 Final evaluation: session 24
  These interventions include: Therapeutic exercises, Perineal electromyographic biofeedback, and Electrical stimulation
  Interventions: Behavioral: Therapeutic exercises; Device: Perineal electromyographic biofeedback; Device: Electrical stimulation
- Premature Ejaculation + Erectile Dysfunction (Experimental): Pelvic Floor Physiotherapy assessment: session 1 Proprioceptive and Coordination Work: sessions 2-12 Muscle workout: sessions 13-20 Functional training: sessions 20-23 Final evaluation: session 24
  These interventions include: Therapeutic exercises, Perineal electromyographic biofeedback, and Electrical stimulation
  Interventions: Behavioral: Therapeutic exercises; Device: Perineal electromyographic biofeedback; Device: Electrical stimulation

INTERVENTIONS:
Behavioral: Therapeutic exercises — Recognition of the pelvic area, respiratory management, lumbo-pelvic mobilization, discrimination of abdomino-pelvic contraction and myofascial release techniques.
Device: Perineal electromyographic biofeedback — Free muscle work and gross motor coordination:
Device: Electrical stimulation — Muscular proprioceptive work: 50 Hz 300 µs

SUMMARY:
The objective of this clinical trial is to evaluate the effectiveness of pelvic floor therapy for the management of erectile dysfunction and premature ejaculation in patients with erectile dysfunction and premature ejaculation. The main question to answer is:

What is the effectiveness of pelvic floor therapy (electrostimulation, biofeedback, and therapeutic exercise) for the treatment of patients with erectile dysfunction and or premature ejaculation?

Patients will:

* Have an initial consultation of pelvic floor rehabilitation before therapy.
* Be given pelvic floor therapy.
* Have a secondary consultation of pelvic floor rehabilitation after therapy.

Three intervention groups will be included: Group 1: Patients with premature ejaculation Group 2: Patients with erectile dysfunction Group 3: Patients with erectile dysfunction and premature ejaculation.

DETAILED DESCRIPTION:
The objective of this clinical trial is to evaluate the effectiveness of pelvic floor therapy for the management of erectile dysfunction and premature ejaculation in patients with erectile dysfunction and premature ejaculation.

Methodology: Pre-post study. Erectile function or intravaginal latency time will be evaluated before and after pelvic floor therapy, in three groups of patients, independently:

* Group 1: Patients with premature ejaculation
* Group 2: Patients with erectile dysfunction
* Group 3: Patients with erectile dysfunction and premature ejaculation

  66 patients will be included and will receive 24 sessions of pelvic floor therapy during 12 weeks. Outcomes will be evaluated at the end of therapy (12 weeks), 3 and 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

Overall:

* Men over 18 years of age
* Erectile dysfunction or premature ejaculation for at least 6 months
* Sexual activity with a heterosexual partner at least once a week
* Signing of informed consent before the start of the study

For the premature ejaculation group:

* Premature ejaculation according to the International Society of Sexual Medicine (ISSM) criteria
* Premature Ejaculation Diagnosis Tool (PEDT) questionnaire score greater than 11

For the erectile dysfunction group:

* Clinical diagnosis of primary erectile dysfunction
* International Index Erectile Function - Erectile Function domain (IIEF-EF) score less than 26

Exclusion Criteria:

* Pharmacological treatment for erectile dysfunction or premature ejaculation in the last 3 months
* Erection Hardness Score (EHS) greater than 3 for patients with erectile dysfunction
* History of hypogonadism or suspected hypogonadism due to Aging Males Symptoms (AMS) score greater than 36 for patients with erectile dysfunction
* History of pelvic radiotherapy
* Pacemaker or cardiac arrhythmia, epilepsy
* History of spinal cord trauma or spinal surgeries.
* Inability to attend therapies or controls
* Illiteracy or cognitive disability that prevents you from completing the questionnaires
* Psychiatric, psychological disorders, or cognitive deficiencies
* Injuries in the area of application of the therapy
* Active pelvic organ cancer

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline intravaginal latency time (IVLT) | 12 weeks
  Change in baseline intravaginal latency time (IVLT) at the end of therapy. (Groups 1,3)
Change in International Index of Erectile Dysfuntion - Erectile Dysfunction domain (IIEF-EF) score | 12 weeks
  International Index of Erectile Dysfuntion - Erectile Dysfunction domain (IIEF-EF) score change at the end of therapy. (Groups 2,3)

SECONDARY OUTCOMES:
Change in baseline intravaginal latency time (IVLT) at follow-up | 3 and 6 months of follow-up.
  Change in IVLT at 3 and 6 months of follow-up. (Groups 1,3)
Change Premature Ejaculation Perfil (PEP) score | 12 weeks, 3 and 6 months follow-up.
  Change in baseline PEP score at the end of therapy, 3 and 6 months of follow-up. (Groups 1,3)
Change in Premature Ejaculation Diagnosis Tool (PEDT) questionnnaire score | 12 weeks, 3 and 6 months follow-up.
  Change in baseline PEDT questionnaire score at the end of therapy, 3 and 6 months follow-up. (Groups 1,3)
Change Intracavity Assessment | 12 weeks, 3 and 6 months follow-up.
  Change in the parameters of the baseline Intracavity Assessment at the end of therapy, 3 and 6 months follow-up.
Side Effects | 12 weeks, 3 and 6 months follow-up.
  Incidente of side effects related to therapy.
Change in International Index of Erectile Dysfuntion - Erectile Dysfunction domain (IIEF-EF) score at follow-up | 3 and 6 months of follow-up.
  International Index of Erectile Dysfuntion - Erectile Dysfunction domain (IIEF-EF) score change at the 3 and 6 months of follow-up. (Groups 2,3)
Change in Erection Hardness Score (EHS) | 12 weeks, 3 and 6 months of follow-up.
  Increase of 1 point in the baseline EHS at the end of therapy, 3 and 6 months of follow-up. (Groups 2,3)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Amaya, Principal Investigator — Boston Medical Group
Locations (1):
- Boston Medical Group Colombia, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No